CLINICAL TRIAL: NCT05106959
Title: Piloting a Motivational Interviewing Shame-Resilience Training
Acronym: MIST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Jennifer Hettema, Associate Professor, University of New Mexico
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20-059
Record Dates: First submitted 2020-06-23; First posted 2021-11-04 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Shame
Keywords: shame resilience; motivational interviewing; shame

STUDY DESIGN:
Intervention Model Description: Longitudinal single group pilot study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pilot Training (Experimental): In this arm participants will complete a variety of baseline assessments then participate in 15-20 minute conversation based on motivational interviewing principles in which they are trained in shame resilience. Follow-ups will be conducted a month later. Assessments will be repeated and then participants will engage in a qualitative interview regarding the training.
  Interventions: Behavioral: Motivational Interviewing Informed Shame Resilience Training

INTERVENTIONS:
Behavioral: Motivational Interviewing Informed Shame Resilience Training — Shame resilience involves four elements. Understating shame, normalizing shame thoughts, reaching out, and speaking shame. Motivational interviewing will be used to elicit and guide participants through these four elements.

SUMMARY:
The purpose of this study is to evaluate the shame resilience theory in a pilot context to assess its feasibility in a potential full scale clinical trial. Shame resilience was developed through qualitative methods but currently has little quantitative backing. Continued research is needed to assess shame-resilience as a potential intervention for shame which little is known to combat prevalent negative health outcomes associated with shame.

DETAILED DESCRIPTION:
Shame is an emotion that can have significant negative impacts on health outcomes, including engagement in care. Feelings of shame are commonly experienced with stigmatized behaviors, such as substance misuse, and may be particularly strong among pregnant women who misuse substances. Rates of opioid misuse during pregnancy are dramatically rising, particularly in New Mexico, leading to negative health outcomes for mothers and fetuses. Shame has been found to decrease these patients' willingness to attend and engage in care. Although a theoretical model is available to guide interventions to reduce shame, it has not been tested empirically. In the current study, investigators seek to evaluate the preliminary effectiveness and feasibility of a brief Shame Resilience Intervention among women seeking care in UNM's Milagro program, a prenatal medical clinic for opioid using pregnant women. This research has the potential to significantly improve public health by generating a tool to reduce barriers to care.

ELIGIBILITY:
Inclusion Criteria:

* Study participants will be Milagro patients
* Engaged in medication assisted treatment
* At least 18 years of age
* Can read and speak English
* Are willing to be contacted for follow-up \
* Are not incarcerated
* Are within the first or second trimester of pregnancy

Exclusion Criteria:

* The study will not enroll non-English speaking Milagro patients
* Patients with obvious cognitive impairments
* Patients with the inability to provide informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-06-26 (Actual); Primary Completion 2020-12-16 (Actual); Study Completion 2021-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Hettema, PhD, Principal Investigator — University of New Mexico Department of Family and Community Medicine
Locations (1):
- South-East Heights Clinic, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No
We currently don't have an IPD sharing plan.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No enrolled participants were excluded from the study
Period: Overall Study
Arm/Group | Pilot Training
Started | 20
Completed | 19
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Pregnant women in first or second trimester with opioid use disorder
Arm/Group | Pilot Training
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: Years] | 29.19 [21 to 39]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 12
  More than one race | 0
  Unknown or Not Reported | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Willingness to Communicate
Description: This measure looks at participants willingness to communicate about their health on a 5 point Likert Scale; 1-5 with higher scores indicating a greater willingness to communicate. Participants respond to a series of questions on a questionnaire.
Time Frame: 1-month
Population: Pregnant women in first or second trimester with opioid use disorder
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pilot Training
Number analyzed (Participants) | 19
score on a scale | 3.3 (.5132)

2. Primary Outcome: Adult Trauma Symptom Checklist
Description: This measure looks at current symptoms of past trauma experiences on a 4 point Likert scale; 0-3 with higher scores indicating a greater presence of adult trauma symptoms. Participants respond to a questionnaire.
Time Frame: 1-month
Population: Pregnant women in first or second trimester with opioid use disorder
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pilot Training
Number analyzed (Participants) | 19
score on a scale | .913 (.6318)

3. Primary Outcome: Shame Compass
Description: This measure looks at the intensity and frequency of shame experiences on a 4 point Likert Scale; 0-3 with higher scores indicating a greater intensity and frequency of shame experiences. Participants respond to a questionnaire.
Time Frame: 1 month
Population: Pregnant women in first or second trimester with opioid use disorder
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pilot Training
Number analyzed (Participants) | 19
score on a scale | 1.54 (.976)

4. Primary Outcome: WHO Big 5 Subjective Well-Being
Description: This measure looks at participants well-being over the past two weeks on a 6 point Likert Scale; 0-5. Scores range from a minimum of 0 to a maximum of 25, with higher scores indicating a better subjective well-being. Participants respond to a questionnaire.
Time Frame: 1-month
Population: Pregnant women in first or second trimester with opioid use disorder
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pilot Training
Number analyzed (Participants) | 19
score on a scale | 15.26 (5.46)

5. Primary Outcome: Shame Resilience Amongst Mental Health Trainees
Description: This measure looks at how much a participant is practicing shame resilience on a 4 point Likert Scale; 0-3 with higher scores indicating better shame resilience. Participants respond to a questionnaire.
Time Frame: 1-month
Population: Pregnant women in first or second trimester with opioid use disorder
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pilot Training
Number analyzed (Participants) | 19
score on a scale | 1.83 (.40)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over a period of one-month. Participants completed one follow-up visit after baseline at one-month intervals.
Arm/Group | Pilot Training
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

LIMITATIONS AND CAVEATS:
Utilizing more than one study-interventionist could potentially have indicated differential outcomes in the administration of the intervention. Finally the study was designed pre-covid and had to be adapted for covid limitations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-28): https://cdn.clinicaltrials.gov/large-docs/59/NCT05106959/Prot_SAP_000.pdf